CLINICAL TRIAL: NCT07365787
Title: Effectiveness of Internet-Based Group Cognitive Behaviour Therapy (GCBT) for Anxiety and Depression Among International Students Studying in Malaysia: A Randomized Controlled Trial
Brief Title: Internet-Based Group CBT for Anxiety and Depression Among International Students
Acronym: DARE Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Shamsa Riaz, PhD Candidate, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JKEUPM-2025-330
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Anxiety and Depression; Internet-based Group Cognitive Behaviour Therapy; Internet-based Group CBT; Internet-based Group CBT Intervention; iGCBT; Internet-based GCBT; International Students; University Students
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be provided with 4 weeks intervention, one hour each, followed by one booster session at 1 month post-intervention.
  Interventions: Behavioral: DARE-Depression and Anxiety Regulation Program
- Waitlist Control Group (No Intervention): The waitlist control group will be provided with 4 weeks intervention, one hour each, followed by one booster session at 1 month post-intervention.

INTERVENTIONS:
Behavioral: DARE-Depression and Anxiety Regulation Program — Participants assigned to this intervention will receive a structured, manual-based online GCCBT intervention delivered via Zoom. The program consists of four weekly group sessions, each lasting approximately 60 minutes, followed by a booster session conducted one month after completion of the intervention.
  Sessions will be conducted by the researcher, a clinical psychologist, under the supervision of a senior clinical psychologist with formal training and expertise in group Cognitive Behavioral Therapy (GCBT). The intervention follows a structured progression beginning with psychoeducation, followed by cognitive skill development and behavioural techniques. The later sessions emphasise consolidation of learnt skills, peer support, and relapse-prevention planning.
  The content and delivery of the intervention are designed to be relevant and sensitive to the experiences of international university students.
  Arms: Experimental Group

SUMMARY:
The goal of this RCT trial is to learn if internet-based group cognitive behaviour therapy delivered via the Zoom application works to treat anxiety and depression among international students. It will also learn about the predictive factors of the intervention's effectiveness. The main questions it aims to answer are:

* Does participating in internet-based GCBT reduce the symptoms of anxiety among international students in Malaysia?
* Does participating in internet-based GCBT reduce the symptoms of depression among international students in Malaysia?

Researchers will compare students who take part in the intervention program with students in a waitlist control group to understand whether the intervention is associated with changes in anxiety and depression symptoms.

Participants will:

* Be randomly assigned to either the intervention program or a waitlist control group
* Attend four sessions of one hour each, including 1) psychoeducation, 2) cognitive techniques, 3) behaviour techniques, and 4) support and relapse prevention. A booster session and a follow-up assessment will be done1 month post intervention.

ELIGIBILITY:
Inclusion Criteria:

* International students.
* 18 and 60 years of age.
* Moderate to severe symptoms of anxiety and depression.
* Fluent in the English language.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale | Baseline, post-intervention at 1 month, and follow-up at one month post-intervention.
  The GAD-7 is a 7-item self-report measure used to assess the frequency and severity of anxiety symptoms in clients 11 and older. Aligned with the DSM-V-TR criteria for Generalized Anxiety Disorder (GAD) the results of this measure can support accurate diagnoses, establishment of treatment goals based on symptom severity, and guide effective clinical interventions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
  Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%) and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
Patient Health Questionnaire | Baseline, post-intervention at 1 month, and follow-up at one month post-intervention.
  The PHQ-9 is a widely recognized self-report questionnaire used to screen for depression severity. It's a simple yet powerful tool, comprising nine questions that mirror the nine diagnostic criteria for major depressive disorder from the DSM-IV. Understanding how to score phq 9 is the first step in interpreting your results.
  A score of ≥10 is considered a sensitive and specific cut-off for major depressive disorder. Whereas, a score ≥15 strongly indicates the presence of clinically significant depression.
Automatic Thoughts Questionnaire | Baseline, post-intervention at 1 month, and follow-up at one month post-intervention.
  The ATQ is a psychological assessment tool designed to measure the frequency of negative automatic thoughts, particularly in individuals with depression.
  ATQ consists of 30 items, each describing a common negative automatic thought relevant to depression, such as "I am a failure" or "I can't cope." Respondents rate how frequently they have experienced each thought over a specified period, typically the past week, using a structured Likert scale. This systematic approach transforms fleeting internal experiences into quantifiable data points.

SECONDARY OUTCOMES:
World Health Organization Quality of Life-BREF | Baseline, post-intervention at 1 month, and follow-up at one month post-intervention.
  WHOQOL-BREF is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health.
  Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. Subsequently, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score, with a higher score indicating a higher QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Firdaus Mukhtar, Study Chair — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia (UPM), Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) will not be shared publicly at this stage. The study is part of a doctoral research project, and data access is restricted to the primary research team to protect participant confidentiality and comply with institutional ethics approval. Any future data sharing would require additional ethical clearance and participant consent.

REFERENCES:
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Hollon, S. D., & Kendall, P. C. (1980). Cognitive self-statements in depression: Development of an automatic thoughts questionnaire. Cognitive Therapy and Research, 4(4), 383-395. https://doi.org/10.1007/BF01178214
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171